CLINICAL TRIAL: NCT06705361
Title: Effect of Ice-Bag Pressure, Transparent Radial Artery (TR) Band Compression Device-Screw, and Air Types on Early Complications and Patient Comfort After Radial Arterial Line Removal in Open Heart Surgery: A Randomized Clinical Trial
Brief Title: Ice Bag, TR Band, and Air Compression Effects on Radial Line Removal Outcomes in Open Heart Surgery: A Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Collaborators: Personalis Inc. (Industry)
Responsible Party: Principal Investigator, Ali Abdul-Rasool Abbas, Master student, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UOB. CON. 24. 002
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Cardiac Disease
Keywords: Ice-bag, TR band device, RA. line removal, Open heart
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transparent Radial Band Compression Device (Screw-Type) (Experimental): To perform TR Band Compression Device (Screw Type) placement after radial arterial line removal, position the patient with the forearm and wrist exposed, ensuring privacy. Place an absorbent pad under the area and clean the puncture site with povidone. Withdraw the radial arterial line by 2-3 cm and secure the TR Band Compression Device with the strap, ensuring it is tight enough to prevent spinning. Adjust the screw cap to control pressure, gradually removing the line while maintaining hemostasis. Use the reverse Barbeau's test to confirm radial artery patency and adjust pressure as needed. After bleeding stops, unfasten the band while stabilizing the site, clean any blood, and apply a sterile gauze dressing. Reassess hand perfusion to ensure adequate blood flow.
  Interventions: Device: Transparent Radial Artery Band (Screw-Type)
- Transparent Radial Band Compression Device (Air-Type) (Experimental): To perform TR Band Compression Device (Air Type) placement after radial arterial line removal, position the patient with the forearm and wrist exposed, ensuring privacy. Place an absorbent pad under the area and clean the puncture site with povidone. Withdraw the radial arterial line by 2-3 cm and secure the TR Band with the strap, aligning the green marker 1-2 mm proximal to the puncture site. Inflate the balloon with 15-18 mL of air using the syringe, removing the arterial line as the balloon inflates. Titrate air by removing 1 mL per minute while monitoring for bleeding or deflate in one step. Use the reverse Barbeau's test to confirm radial artery patency and adjust air volume as needed. Once hemostasis is achieved, deflate the band, unfasten it, clean the site, and apply a sterile gauze dressing. Reassess hand perfusion to ensure adequate blood flow.
  Interventions: Device: Transparent Radial Artery Band (Screw-Type)
- Ice-Bag Pressure (Experimental): Titrate pressure using the TR Band's mechanical screw cap to maintain patent hemostasis. If bleeding occurs during pressure release, restore compression. Confirm radial pulse and evaluate artery patency using the reverse Barbeau's test. Place an oxygen saturation probe on the thumb or index finger and compress the ulnar artery, observing the waveform. If absent, reduce pressure until the waveform returns, ensuring antegrade flow. Once pressure is fully released, confirm bleeding has stopped. Stabilize the access site, unfasten, and remove the band slowly. Clean any blood with sterile gauze, apply a dressing (not encircling the wrist), and reassess hand perfusion. Ensure proper positioning for left or right wrist use.
  Interventions: Device: Transparent Radial Artery Band (Screw-Type)

INTERVENTIONS:
Device: Transparent Radial Artery Band (Screw-Type) — The researcher will randomly assign patients undergoing radial arterial line removal after open heart surgery into four groups: ice-bag pressure, transparent radial band compression device (screw type), transparent radial band compression device (air type), and control group. The researcher will assign specific card colors to each group: white for the control group, yellow for the ice-bag pressure group, pink for the Transparent Radial Band Compression Device - Screw Type group, and green for the Transparent Radial Band Compression Device - Air Type group. The researcher will place all these cards in a container, allowing the participant to select their preferred color, and then apply the intervention separately to each group.
  Other Names: Transparent Radial Artery Band (Air-Type); Ice-Bag Pressure

SUMMARY:
The study aims to find the different effects of applying an ice-bag pressure, TR radial band compression device-screw type, and TR radial band compression device-air type on early complications and comfort among patients undergoing radial arterial line removal after open heart surgery.

DETAILED DESCRIPTION:
This study will be designed as a randomized control trial (RCT). A randomized controlled trial (RCT) is a research method that encompasses prospective, comparative, quantitative, genuine experimental, and post-test-only control group designs. This type of design will conduct under controlled conditions which allows the researcher to assigned interventions randomly to different groups in order to minimize bias and understand the best cause-and-effect relationship between independent variables (Ice-bag pressure, TR radial band compression device-screw type, and TR radial band compression device-air type) and dependent variables (early complication; bleeding severity, hematoma formation, and patient comfort), as well as this study will utilize the effect of an ice-bag pressure, TR radial band compression device-screw type, and TR radial band compression device-air type as interventions to measure their effectiveness in the reducing of early complication; bleeding severity, hematoma formation, and patient comfort following to radial arterial line removal after open heart surgery and which intervention is more effective. Each individual participating in this study will have an equal chance of being assigned to either the experimental or control group.

Setting:

The research will be carried out at the Ibn Al-Bitar center for cardiac surgery, which has five rooms dedicated to open heart surgery, twelve beds for the postoperative cardiac intensive care unit (CICU), and four beds for the high dependency unit (HDU). Additionally, the Iraqi center for heart disease will be used, which has three rooms for open heart surgery, five beds for post-operative cardiac intensive care unit (CICU), and three beds for high dependency unit (HDU). Situated in the Baghdad governorate, this is a government-operated specialized facility dedicated to open heart surgery and cardiac catheterization. The facilities consistently carry out surgical procedures on approximately 3 cases per day, 15 cases per week, 60 cases per month, and over 720 cases per year, along with emergency operations following a predetermined schedule. This allows for reliable evaluation of the administrative feasibility and availability of the study population.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

Eligible male and female patients who are willing to participate and will have their radial artery lines removed after open heart surgery will be chosen based on specific inclusion criteria. The requirements are as follows: the patient must be at least eighteen years old, orientated, free of visual or auditory impairments, able to communicate orally in Arabic, having a radial intervention which include the insertion of a single arterial line in the radial region, and not taken analgesics for a minimum of three hours.

Exclusion Criteria:

* Exclusion criteria:

The study's exclusion criteria include patients who are unable to communicate due to visual impairment or hearing impairment, as effective communication is essential for data gathering; patients with cognitive disorders; patients experiencing hemodynamic instability, as the implementation of the program necessitates patient compliance; patients with bleeding and hematoma in the radial artery region before arterial line removal; patients with clotting factor disorders; patients with arterial line cutdown; and patients with a documented history of radial disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-11-25 (Estimated); Primary Completion 2025-02-25 (Estimated); Study Completion 2025-03-25 (Estimated)

PRIMARY OUTCOMES:
To assess the comfort level during the procedure as measured by the Numerical Visual Rating Comfort Scale (NVRC scale). | Baseline, within procedure time
  NVRC scale measures overall comfort on a 0-10 scale as follows: "No comfort" (0), "Negligible comfort" (1), "Moderate comfort" (2), "Moderate comfort" (3), "Moderate comfort" (4), "Moderate comfort" (5), "Moderate and fairly high comfort" (6), "Fairly high comfort" (7), "Very high comfort" (8), "Highest comfort possible" (9), A ruler is used to quantify the distance (0 mm) between the anchor and the mark specified by the client on the NVRC scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Abdul-Rasool Abbas, Student, Principal Investigator — University of Baghdad / College of Nursing
Locations (1):
- Ali Abdul-Rasool Abbas, Karbala, Al-bahadliya, Iraq

IPD SHARING:
Plan to Share IPD: No